CLINICAL TRIAL: NCT01820572
Title: Evaluation of the Benefits and Risks in Maintenance Renal Transplant Recipients Following Conversion to Nulojix® (Belatacept)-Based Immunosuppression
Brief Title: A Study in Maintenance Kidney Transplant Recipients Following Conversion to Nulojix® (Belatacept)-Based
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM103-116; 2012-001314-42 (EudraCT Number)
Record Dates: First submitted 2013-03-14; First posted 2013-03-29 (Estimated); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Abatacept; Tacrolimus; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Belatacept (Experimental): Belatacept 5 mg/kg intravenous 30 minute infusion on Days 1, 15, 29, 43, 57 then every 28 days for 24 months
  Interventions: Drug: Belatacept
- CNI (Active Comparator): Tacrolimus 4-11 ng/mL tablet orally according to package insert for 24 months
  Cyclosporine 50-250 ng/mL tablet orally according to package insert for 24 months
  Interventions: Drug: Tacrolimus; Drug: Cyclosporine

INTERVENTIONS:
Drug: Belatacept
  Other Names: BMS 224818; Nulojix®
  Arms: Belatacept
Drug: Tacrolimus
  Arms: CNI
Drug: Cyclosporine
  Arms: CNI

SUMMARY:
The primary purpose is to assess the benefits and risks of changing from Cyclosporine or Tacrolimus to Belatacept between 6-60 months after kidney transplant.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Men and women, ages 18-75 inclusive
* Adult recipients of a renal allograft from a living donor or a deceased donor between 6-60 months prior to enrollment
* Receiving a stable (≥1 month) regimen of Calcineurin inhibitor (CNI) [Cyclosporine A (CsA) or Tacrolimus (TAC)] with Mycophenolate mofetil (MMF) or Enteric Coated Mycophenolate Sodium (EC-MPS)/Mycophenolic acid (MPA), and corticosteroids
* Stable renal function for 12 weeks prior to enrollment without new onset proteinuria
* Calculated glomerular filtration rate (cGFR) ≥30 and ≤75 mL/min/1.73 m2 [Modification of Diet in Renal Disease study (MDRD) 4-formula]

Exclusion Criteria:

* Recipients with Epstein-Barr virus (EBV) serostatus negative or unknown
* History of acute rejection (AR) within 3 months prior to enrollment
* History of antibody mediated rejection
* Positive T-cell lymphocytotoxic cross match
* Proteinuria >1 g/day or >0.5 g/day if diabetic

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 446 (Actual)
Dates: Start 2013-03-27 (Actual); Primary Completion 2019-10-24 (Actual); Study Completion 2019-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (114):
- United States (60):
  - UAB Division of Nephrology, Birmingham, Alabama
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Loma Linda University Medical Center (LLUMC) - Children's Hospital - Transplantation Institute, Loma Linda, California
  - UCLA Kidney Transplant Research Office, Los Angeles, California
  - Keck Medical Center of USC (PI Address), Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Transplant Research Institute (PI Address), Los Angeles, California
  - University of California, San Francisco (UCSF)-Kidney Transplant Service, Sacramento, California
  - California Institute Of Renal Research, San Diego, California
  - California Pacific Medical Center, Depart of Transplantation (PI Address), San Francisco, California
  - UCSF Medical Center, San Francisco, California
  - University of Colorado Denver (PI Address), Aurora, Colorado
  - Denver Nephrologists, PC, Denver, Colorado
  - Yale Medical Group, New Haven, Connecticut
  - Florida Hospital Transplant Institute (PI Address), Orlando, Florida
  - Central Pharmacy, St. Petersburg, Florida
  - Tampa General Medicine Group, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Medical College of Georgia at Augusta University, Augusta, Georgia
  - RUSH University Transplant Program (PI Address), Chicago, Illinois
  - University of Wisconsin School of Medicine and Public Health (PI Address), Chicago, Illinois
  - University of Iowa Health Care (PI Address), Iowa City, Iowa
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Maine Transplant Program, Portland, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Henry Ford's Transplant Institute, Detroit, Michigan
  - St. Clair Nephrology Research, Roseville, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington Univ School of Med, St Louis, Missouri
  - University or Nebraska Medical Center, Omaha, Nebraska
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - University of Buffalo, Buffalo, New York
  - Recanati/Miller Transplantation Institue (PI Address), New York, New York
  - Carolinas Medical Center (PI Address), Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina Univ Nephrology Clin Res. Lab, Greenville, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Central PA Transplant Foundation, Harrisburg, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Penn Medicine, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, SCTR Research Nexus, Charleston, South Carolina
  - Methodist University Hospital Transplant Institute (PI Address), Memphis, Tennessee
  - Vanderbilt University Medical Center- GI Research Office, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor All Saints Medical Center at Ft. Worth, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Memorial Hermann - Texas Medical Center (Tmc), The University Of Texas Medical School At Houston, Houston, Texas
  - The Methodist Hospital, Houston, Texas
  - University of Utah Depart of Nephrology (PI Address), Salt Lake City, Utah
  - University of Virginia Health System (PI Address), Charlottesville, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Virginia Commonwealth University Medical Center, Richmond, Virginia
  - Swedish Medical Center-Swedish Organ Transplant and Liver Center, Seattle, Washington
  - University of Washington Medical Center (PI Address & Study Supplies Address), Seattle, Washington
  - Providence Sacred Heart Medical Center and Childrens Hospital, Spokane, Washington
  - Medical College of WI Froedtert Hospital, Milwaukee, Wisconsin
- Argentina (8):
  - Local Institution, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Local Institution, Mendoza, Buenos Aires
  - Local Institution, Cardoba, Córdoba Province
  - Local Institution, Rosario, Santa Fe Province
  - Local Institution, Buenos Aires
  - Local Institution, CABA
  - Local Institution, Córdoba
  - Local Institution, Santa Fe
- Austria (5):
  - Local Institution, Feldkirch
  - Local Institution, Graz
  - Local Institution, Innsbruck
  - Local Institution, Linz
  - Local Institution, Vienna
- Colombia (2):
  - Local Institution, Cali, Valle del Cauca Department
  - Local Institution, Bogotá
- France (11):
  - Local Institution, Paris, Cedex 15
  - Local Institution, Bois-Guillaume
  - Local Institution, Bordeaux
  - Local Institution, Brest
  - Local Institution, Créteil
  - Local Institution, Grenoble
  - Local Institution, Le Kremilin Bicretre
  - Local Institution, Lyon
  - Local Institution, Paris
  - Local Institution, Strasbourg
  - CHU Rangueil, Toulouse
- Germany (15):
  - Local Institution, Berlin
  - Local Institution, Dresden
  - Local Institution, Erlangen
  - Local Institution, Essen
  - Local Institution, Frankfurt am Main
  - Local Institution, Hamburg
  - Local Institution, Hanover
  - Local Institution, Heidelberg
  - Local Institution, Kiel
  - Local Institution, Lübeck
  - Local Institution, Mannheim
  - Local Institution, München
  - Local Institution, Münster
  - Local Institution, Regensburg
  - Local Institution, Würzburg
- Netherlands (5):
  - Local Institution, Amsterdam
  - Local Institution, Groningen
  - Local Institution, Leiden
  - Local Institution, Nijmegen
  - Local Institution, Utrecht
- Norway (2):
  - Local Institution, Oslo
  - Local Institution, Toensberg Norge
- Sweden (3):
  - Local Institution, Gothenburg
  - Local Institution, Stockholm
  - Local Institution, Uppsala
- Switzerland (3):
  - Local Institution, Bern
  - Local Institution, Geneva
  - Local Institution, Zurich

REFERENCES:
- [Derived] Budde K, Prashar R, Haller H, Rial MC, Kamar N, Agarwal A, de Fijter JW, Rostaing L, Berger SP, Djamali A, Leca N, Allamassey L, Gao S, Polinsky M, Vincenti F. Conversion from Calcineurin Inhibitor- to Belatacept-Based Maintenance Immunosuppression in Renal Transplant Recipients: A Randomized Phase 3b Trial. J Am Soc Nephrol. 2021 Dec 1;32(12):3252-3264. doi: 10.1681/ASN.2021050628. Epub 2021 Dec 1. PMID 34706967
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 446 Enrolled and Treated
Groups:
- Belatacept: Participants who converted to belatacept treatment from CNI-Based
- CNI-Based Regimen: Participants who continued on CNI-Based regimens
Period: Randomization
Arm/Group | Belatacept | CNI-Based Regimen
Started (= Participants Randomized) | 223 | 223
Completed (= Participants Treated) | 221 | 222
Not Completed | 2 | 1
Not completed — Not Treated | 2 | 1
Period: Treatment Period
Arm/Group | Belatacept | CNI-Based Regimen
Started (= participants treated) | 221 | 222
Completed (= participants completing treatment) | 195 | 186
Not Completed | 26 | 36
Not completed — Adverse Event | 12 | 7
Not completed — Death | 3 | 3
Not completed — Lack of Efficacy | 1 | 0
Not completed — poor/non compliance | 0 | 3
Not completed — request to discontinue | 6 | 11
Not completed — No longer meets study criteria | 3 | 10
Not completed — withdrew consent | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Belatacept | CNI-Based Regimen | Total
Number analyzed (Participants) | 223 | 223 | 446
Age, Continuous [Median (Standard Deviation); unit: Years] | 55.0 (11.3) | 54.0 (11.7) | 54.0 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 72 | 145
  Male | 150 | 151 | 301
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 15 | 24
  Not Hispanic or Latino | 82 | 79 | 161
  Unknown or Not Reported | 132 | 129 | 261
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 24 | 24 | 48
  White | 191 | 187 | 378
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 9 | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Survive With a Functional Graft at 24 Months
Description: Percentage of participants who survive with a functional graft at 24 months post-randomization
Time Frame: at 24 Months
Population: All Randomized Participants
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Belatacept | CNI-Based Regimen
Number analyzed (Participants) | 223 | 223
Percentage | 98.2 [95.5 to 99.5] | 97.3 [95.2 to 99.4]
Statistical Analysis 1: Comparison: Belatacept vs CNI-Based Regimen; Test type: Superiority — difference between belatacept and CNI; Difference in proportions = 0.9, 95% CI 2-sided [-8.6 to 10.4]

2. Secondary Outcome: Percentage of Participants Who Survive With a Functional Graft at 12 Months
Description: Percentage of participants who survive with a functional graft at 12 months post-randomization
Time Frame: at 12 Months
Population: All Randomized Participants
Measure: Number (95% Confidence Interval); unit: Percentage
Arm/Group | Belatacept | CNI-Based Regimen
Number analyzed (Participants) | 223 | 223
Percentage | 98.7 [96.1 to 99.7] | 99.1 [96.8 to 99.9]
Statistical Analysis 1: Comparison: Belatacept vs CNI-Based Regimen; Test type: Superiority — difference between belatacept and CNI; Difference in Proportions = -0.4, 95% CI 2-sided [-9.9 to 9.0]

3. Secondary Outcome: Number of Participants With a Biopsy Proven Acute Rejection (BPAR)
Description: The number of clinically suspected, biopsy proven acute rejection (AR) at 12 and 24 months post-randomization
  includes participants with at least one cellular and/or humoral BPAR event.
Time Frame: at 12 and 24 Months
Population: All Randomized Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Belatacept | CNI-Based Regimen
Number analyzed (Participants) | 223 | 223
Participants
  at 12 Months | 18 | 4
  at 24 Months | 18 | 9

4. Secondary Outcome: Number of Participants With Varying Severity of BPAR
Description: Number of participants in each severity of clinically suspected, biopsy proven acute rejection (AR) at 12 and 24 months post-randomization
Time Frame: at 12 and 24 months
Population: All Randomized Participants who had a BPAR
Measure: Count of Participants; unit: Participants
Arm/Group | Belatacept | CNI-Based Regimen
Number analyzed (Participants) | 20 | 6
Participants
  at 12 Months: number analyzed (Participants) | 20 | 3
  at 12 Months: Mild Acute (IA) | 2 | 2
  at 12 Months: Mild Acute (IB)1 | 1 | 0
  at 12 Months: Moderate Acute (IIA) | 7 | 0
  at 12 Months: Moderate Acute (IIB) | 6 | 0
  at 12 Months: Severe Acute (III) | 4 | 1
  at 24 Months: Mild Acute (IA) | 2 | 4
  at 24 Months: Mild Acute (IB)1 | 1 | 0
  at 24 Months: Moderate Acute (IIA) | 7 | 1
  at 24 Months: Moderate Acute (IIB) | 6 | 0
  at 24 Months: Severe Acute (III) | 4 | 1

5. Secondary Outcome: Mean Change From Baseline of Calculated Glomerular Filtration Rate (cGFR) - Percent Change
Description: Mean change from baseline cGFR as calculated by the 4-variable MDRD equation to 12 and 24 months post-randomization - Percent Change
Time Frame: at 12 and 24 months
Population: All Randomized Participants
Measure: Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Belatacept | CNI-Based Regimen
Number analyzed (Participants) | 223 | 223
Percent Change
  at 12 Months: number analyzed (Participants) | 196 | 190
  at 12 Months | 13.2 [10.4 to 16.0] | -0.3 [-2.9 to 2.4]
  at 24 Months: number analyzed (Participants) | 189 | 171
  at 24 Months | 15.2 [11.9 to 18.6] | 0.3 [-2.9 to 3.4]

6. Secondary Outcome: Mean Change From Baseline of Calculated Glomerular Filtration Rate (cGFR) - Adjusted Change
Description: Mean change from baseline cGFR as calculated by the 4-variable MDRD equation to 12 and 24 months post-randomization - Adjusted Change
Time Frame: at 12 and 24 months
Population: All Randomized Participants
Measure: Mean (95% Confidence Interval); unit: mL/min/1.73m²
Arm/Group | Belatacept | CNI-Based Regimen
Number analyzed (Participants) | 223 | 223
mL/min/1.73m²
  at 12 Months | 5.6 [4.3 to 6.9] | -0.7 [-2.0 to 0.6]
  at 24 Months | 6.2 [4.7 to 7.7] | -1.0 [-2.6 to 0.5]

7. Secondary Outcome: Mean Calculated Glomerular Filtration Rate (cGFR)
Description: Mean cGFR by study visit, as calculated by the 4-variable MDRD equation.
Time Frame: up to 24 months
Population: All Randomized Participants
Measure: Mean (95% Confidence Interval); unit: mL/min/1.73m²
Arm/Group | Belatacept | CNI-Based Regimen
Number analyzed (Participants) | 223 | 223
mL/min/1.73m²
  Screening | 49.8 [48.2 to 51.5] | 49.7 [48.2 to 51.2]
  Baseline | 49.6 [48.0 to 51.2] | 50.7 [49.2 to 52.2]
  Month 3: number analyzed (Participants) | 215 | 206
  Month 3 | 53.0 [51.1 to 54.9] | 50.2 [48.3 to 52.0]
  Month 6: number analyzed (Participants) | 200 | 199
  Month 6 | 53.3 [51.3 to 55.3] | 50.9 [49.1 to 52.7]
  Month 9: number analyzed (Participants) | 195 | 182
  Month 9 | 53.7 [51.8 to 55.6] | 50.7 [48.9 to 52.5]
  Month 12: number analyzed (Participants) | 196 | 190
  Month 12 | 55.5 [53.4 to 57.6] | 50.5 [48.7 to 52.4]
  Month 18: number analyzed (Participants) | 185 | 173
  Month 18 | 56.5 [54.5 to 58.5] | 51.3 [49.2 to 53.4]
  Month 24: number analyzed (Participants) | 189 | 171
  Month 24 | 55.7 [53.7 to 57.7] | 51.1 [49.0 to 53.2]

8. Secondary Outcome: Slope Analysis of cGFR
Description: Slopes of cGFR as plotted from baseline as well as from Month 3, to Month 12 and Month 24 post-randomization
Time Frame: at 12 and 24 Months
Population: All Randomized Participants
Measure: Number (95% Confidence Interval); unit: mL/min/1.73m²/month
Arm/Group | Belatacept | CNI-Based Regimen
Number analyzed (Participants) | 223 | 223
mL/min/1.73m²/month
  Baseline to 12 Months | 0.241 [0.103 to 0.378] | 0.004 [-0.137 to 0.145]
  Month 3 to Month 12 | 0.281 [0.072 to 0.490] | -0.159 [-0.372 to 0.055]
  Baseline to Month 24 | 0.685 [0.426 to 0.945] | -0.112 [-0.379 to 0.155]
  Month 3 to Month 24 | 0.658 [0.332 to 0.984] | -0.277 [-0.614 to 0.060]

9. Secondary Outcome: Slope Analysis of 1/Serum Creatinine
Description: Slopes of 1/serum creatinine as plotted from baseline as well as from Month 3, to Month 12 and Month 24 post-randomization
Time Frame: at 12 and 24 Months
Population: All Randomized Participants
Measure: Number (95% Confidence Interval); unit: mg/dL/month
Arm/Group | Belatacept | CNI-Based Regimen
Number analyzed (Participants) | 223 | 223
mg/dL/month
  Baseline to 12 Months | 0.034 [0.016 to 0.051] | -0.003 [-0.020 to 0.015]
  Month 3 to Month 12 | 0.033 [0.007 to 0.059] | -0.021 [-0.048 to 0.006]
  Baseline to Month 24 | 0.00868 [0.00537 to 0.01199] | -0.00203 [-0.00544 to 0.00138]
  Month 3 to Month 24 | 0.00814 [0.00412 to 0.01217] | -0.00425 [-0.00842 to -0.00009]

10. Secondary Outcome: Percentage of Participants With > 5% and >10% Improvement Over Baseline cGFR
Description: Percentage of participants with > 5% and >10% improvement over baseline cGFR, at 12 and 24 months post-randomization
Time Frame: at 12 and 24 Months
Population: All Randomized Participants
Measure: Number; unit: Percentage
Arm/Group | Belatacept | CNI-Based Regimen
Number analyzed (Participants) | 223 | 223
Percentage
  >5% improvement at 12 months: number analyzed (Participants) | 119 | 64
  >5% improvement at 12 months | 53.4 | 28.7
  >10% improvement at 12 months: number analyzed (Participants) | 98 | 48
  >10% improvement at 12 months | 43.9 | 21.5
  >5% improvement at 24 months: number analyzed (Participants) | 121 | 66
  >5% improvement at 24 months | 54.3 | 29.6
  >10% improvement at 24 months: number analyzed (Participants) | 108 | 49
  >10% improvement at 24 months | 48.4 | 22.0

11. Secondary Outcome: Mean Urine Protein/ Creatinine Ratio (UPCR)
Description: Urine protein/ creatinine ratio (UPCR) at baseline, 3, 6, 12 and 24 months post randomization
Time Frame: Up to 24 Months
Population: All Randomized Participants
Measure: Mean (95% Confidence Interval); unit: mg/mmol
Arm/Group | Belatacept | CNI-Based Regimen
Number analyzed (Participants) | 223 | 223
mg/mmol
  at Baseline: number analyzed (Participants) | 222 | 221
  at Baseline | 17.80 [16.03 to 19.58] | 18.61 [15.08 to 22.14]
  at 3 months: number analyzed (Participants) | 204 | 184
  at 3 months | 22.87 [19.88 to 25.86] | 20.61 [15.50 to 25.73]
  at 6 months: number analyzed (Participants) | 196 | 194
  at 6 months | 23.42 [19.71 to 27.12] | 20.85 [15.36 to 26.35]
  at 12 months: number analyzed (Participants) | 189 | 183
  at 12 months | 29.11 [21.86 to 36.35] | 21.67 [17.70 to 25.65]
  at 24 months: number analyzed (Participants) | 188 | 169
  at 24 months | 28.81 [23.71 to 33.91] | 24.56 [19.01 to 30.10]

12. Secondary Outcome: Mean Change From Baseline in Systolic and Diastolic Blood Pressure
Description: Mean change in systolic and diastolic blood pressure from baseline to 12 and 24 months post randomization
Time Frame: at 12 and 24 months
Population: All Randomized Participants
Measure: Mean (90% Confidence Interval); unit: mmHg
Arm/Group | Belatacept | CNI-Based Regimen
Number analyzed (Participants) | 223 | 223
mmHg
  Diastolic BP at 12 Months: number analyzed (Participants) | 198 | 196
  Diastolic BP at 12 Months | -1.5 [-2.9 to 0.0] | -0.6 [-2.1 to 1.0]
  Diastolic BP at 24 Months: number analyzed (Participants) | 193 | 173
  Diastolic BP at 24 Months | -1.7 [-3.3 to 0.0] | 0.5 [-1.3 to 2.3]
  Systolic BP at 12 Months: number analyzed (Participants) | 198 | 196
  Systolic BP at 12 Months | -1.6 [-4.0 to 0.9] | 0.1 [-2.5 to 2.8]
  Systolic BP at 24 Months: number analyzed (Participants) | 193 | 173
  Systolic BP at 24 Months | -1.3 [-4.1 to 1.6] | 1.2 [-1.7 to 4.1]

13. Secondary Outcome: Number of Antihypertensive Medications Used to Control Hypertension
Description: The total number of antihypertensive medications used to control hypertension
Time Frame: at baseline, 12 and 24 Months
Population: All Randomized Participants
Measure: Mean (Full Range); unit: Number of medications
Arm/Group | Belatacept | CNI-Based Regimen
Number analyzed (Participants) | 223 | 223
Number of medications
  at Baseline: number analyzed (Participants) | 195 | 191
  at Baseline | 2.1 [1 to 5] | 2.2 [1 to 6]
  at 12 Months: number analyzed (Participants) | 194 | 195
  at 12 Months | 2.3 [1 to 7] | 2.2 [1 to 6]
  at 24 Months: number analyzed (Participants) | 193 | 190
  at 24 Months | 2.3 [1 to 8] | 2.3 [1 to 7]

14. Secondary Outcome: Number of Participants With Donor Specific Antibodies (DSA)
Description: Number of participants with donor specific antibodies (DSA) at Baseline/Day 1, and Months 12 and 24 post-randomization
Time Frame: at baseline, 12 and 24 months
Population: All Randomized Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Belatacept | CNI-Based Regimen
Number analyzed (Participants) | 223 | 223
Participants
  Pre Existing at baseline: number analyzed (Participants) | 207 | 199
  Pre Existing at baseline | 10 | 26
  De Novo at 12 Months: number analyzed (Participants) | 219 | 216
  De Novo at 12 Months | 2 | 9
  De Novo at 24 Months: number analyzed (Participants) | 221 | 199
  De Novo at 24 Months | 2 | 14

15. Secondary Outcome: Mean Number of Symptom Occurrence and Symptom Distress
Description: The frequency of symptom occurrence and symptom distress as measured with the Modified Transplant Symptom Occurrence and Symptom Distress Scale-59R (MTSOSD-59R) at baseline, Week 6, and Months 3, 6, and 12 post-randomization.
  Higher scores in the MTSOSD-59R indicate a greater symptom and symptom distress burden than lower scores.
Time Frame: up to 12 Months
Population: All randomized and Treated Participants
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Belatacept | CNI-Based Regimen
Number analyzed (Participants) | 223 | 223
Scores on a scale
  Baseline symptom occurrence: number analyzed (Participants) | 212 | 218
  Baseline symptom occurrence | 87.8 (20.06) | 90.7 (21.04)
  Baseline symptom distress: number analyzed (Participants) | 211 | 216
  Baseline symptom distress | 28.7 (27.07) | 34.8 (28.30)
  week 6 symptom occurrence: number analyzed (Participants) | 209 | 193
  week 6 symptom occurrence | 79.0 (16.52) | 88.6 (21.36)
  week 6 symptom distress: number analyzed (Participants) | 204 | 193
  week 6 symptom distress | 19.8 (21.41) | 32.4 (29.55)
  Month 3 symptom occurrence: number analyzed (Participants) | 207 | 196
  Month 3 symptom occurrence | 80.5 (16.74) | 89.9 (23.45)
  Month 3 symptom distress: number analyzed (Participants) | 200 | 194
  Month 3 symptom distress | 21.4 (23.08) | 35.2 (32.04)
  month 6 symptom occurrence: number analyzed (Participants) | 198 | 189
  month 6 symptom occurrence | 80.5 (17.50) | 91.8 (23.72)
  month 6 symptom distress: number analyzed (Participants) | 189 | 185
  month 6 symptom distress | 22.4 (22.18) | 36.3 (31.39)
  month 12 symptom occurrence: number analyzed (Participants) | 196 | 188
  month 12 symptom occurrence | 82.3 (20.08) | 91.0 (22.33)
  month 12 symptom distress: number analyzed (Participants) | 185 | 186
  month 12 symptom distress | 25.8 (25.32) | 34.4 (30.82)

16. Secondary Outcome: Number of Participants With an Adverse Event of Special Interest
Description: Number of participants with an adverse event of special interests. Adverse events of special interest include:
  Serious Infections, Post-Transplant Lymphoproliferative Disorder (PTLD), Progressive multifocal leukoencephalopathy (PML), Malignancies (other than PTLD) including non-melanoma skin carcinomas, Tuberculosis Infections, CNS infections, Viral Infections and Infusion related reactions.
Time Frame: 24 Months
Population: As Treated Population
Measure: Number; unit: participants
Arm/Group | Belatacept | CNI-Based Regimen
Number analyzed (Participants) | 221 | 222
participants
  Serious Infections | 37 | 44
  PTLD | 1 | 0
  PML | 0 | 0
  Malignancies | 17 | 12
  Tuberculosis infections | 0 | 0
  CNS Infections | 0 | 0
  Viral Infections | 5 | 9
  Infusion Related Reactions | 13 | 0

17. Secondary Outcome: Number of Participants With Marked Laboratory Abnormalities
Description: Number of participants with Marked Laboratory Abnormalities
Time Frame: 24 Months
Population: All Randomized and Treated Participants
Measure: Number; unit: Participants
Arm/Group | Belatacept | CNI-Based Regimen
Number analyzed (Participants) | 221 | 222
Participants
  Hemoglobin (Abnormal Low): number analyzed (Participants) | 218 | 212
  Hemoglobin (Abnormal Low) | 0 | 0
  Hemoglobin (Abnormal high): number analyzed (Participants) | 218 | 212
  Hemoglobin (Abnormal high) | 0 | 0
  Platelet count (Abnormal low): number analyzed (Participants) | 218 | 213
  Platelet count (Abnormal low) | 0 | 1
  Leukocytes (Abnormal low): number analyzed (Participants) | 218 | 213
  Leukocytes (Abnormal low) | 0 | 0
  Lymphocytes (Abnormal low): number analyzed (Participants) | 218 | 212
  Lymphocytes (Abnormal low) | 29 | 10
  Lymphocytes (Abnormal high): number analyzed (Participants) | 218 | 212
  Lymphocytes (Abnormal high) | 0 | 0
  Neutrophils Absolute (Abnormal low): number analyzed (Participants) | 218 | 212
  Neutrophils Absolute (Abnormal low) | 5 | 3
  Alanine Aminotransferase (Abnormal High): number analyzed (Participants) | 219 | 213
  Alanine Aminotransferase (Abnormal High) | 0 | 0
  Alkaline Phosphatase (Abnormal High): number analyzed (Participants) | 219 | 213
  Alkaline Phosphatase (Abnormal High) | 0 | 0
  Aspartate Aminotransferase (Abnormal High): number analyzed (Participants) | 219 | 213
  Aspartate Aminotransferase (Abnormal High) | 0 | 1
  Total Bilirubin (Abnormal High): number analyzed (Participants) | 219 | 213
  Total Bilirubin (Abnormal High) | 0 | 0
  Creatine (Abnormal High): number analyzed (Participants) | 220 | 218
  Creatine (Abnormal High) | 5 | 4
  Protein/Creatinine Ratio (Abnormal High): number analyzed (Participants) | 217 | 213
  Protein/Creatinine Ratio (Abnormal High) | 0 | 0
  Bicarbonate (Abnormal High): number analyzed (Participants) | 219 | 213
  Bicarbonate (Abnormal High) | 0 | 1
  Total Calcium (Abnormal low): number analyzed (Participants) | 219 | 213
  Total Calcium (Abnormal low) | 0 | 3
  Total Calcium (Abnormal high): number analyzed (Participants) | 219 | 213
  Total Calcium (Abnormal high) | 1 | 2
  Magnesium (Abnormal low): number analyzed (Participants) | 219 | 213
  Magnesium (Abnormal low) | 0 | 0
  Magnesium (Abnormal high): number analyzed (Participants) | 219 | 213
  Magnesium (Abnormal high) | 0 | 0
  Phosphorus (Abnormal Low): number analyzed (Participants) | 219 | 213
  Phosphorus (Abnormal Low) | 14 | 12
  Potassium (Abnormal low): number analyzed (Participants) | 219 | 213
  Potassium (Abnormal low) | 3 | 2
  Potassium (Abnormal high): number analyzed (Participants) | 219 | 213
  Potassium (Abnormal high) | 1 | 5
  Sodium (Abnormal low): number analyzed (Participants) | 219 | 213
  Sodium (Abnormal low) | 4 | 9
  Sodium (Abnormal high): number analyzed (Participants) | 219 | 213
  Sodium (Abnormal high) | 0 | 1
  Albumin (Abnormal low): number analyzed (Participants) | 219 | 213
  Albumin (Abnormal low) | 0 | 0
  Total Cholesterol (Abnormal High): number analyzed (Participants) | 208 | 205
  Total Cholesterol (Abnormal High) | 13 | 17
  Serum Glucose (Abnormal low): number analyzed (Participants) | 205 | 208
  Serum Glucose (Abnormal low) | 0 | 0
  Serum Glucose (Abnormal high): number analyzed (Participants) | 205 | 208
  Serum Glucose (Abnormal high) | 18 | 18
  Triglycerides (Abnormal high): number analyzed (Participants) | 186 | 188
  Triglycerides (Abnormal high) | 2 | 2
  Uric Acid (Abnormal high): number analyzed (Participants) | 219 | 213
  Uric Acid (Abnormal high) | 15 | 30

18. Secondary Outcome: Mean Change From Baseline in Vital Signs: Heart Rate
Description: The mean change from baseline in measured heart rate
Time Frame: at 12 and 24 months
Population: All Randomized and Treated Participants
Measure: Mean (95% Confidence Interval); unit: beats per minute (bpm)
Arm/Group | Belatacept | CNI-Based Regimen
Number analyzed (Participants) | 221 | 222
beats per minute (bpm)
  Change from baseline at 12 months: number analyzed (Participants) | 197 | 166
  Change from baseline at 12 months | -1.8 [-3.3 to -0.2] | -0.6 [-2.2 to 1.0]
  Change from baseline at 24 months: number analyzed (Participants) | 192 | 149
  Change from baseline at 24 months | -1.9 [-3.5 to -0.3] | 1.0 [-0.8 to 2.8]

ADVERSE EVENTS:
Time Frame: 116 Weeks
Arm/Group | Belatacept | CNI-Based Regimen
All-Cause Mortality (participants affected / at risk) | 4/221 | 5/222
Serious Adverse Events (participants affected / at risk) | 107/221 | 95/222
Other Adverse Events (participants affected / at risk) | 174/221 | 168/222
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Belatacept (N=221) | CNI-Based Regimen (N=222)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 0
Monocytosis (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 3
Coronary artery disease (Cardiac disorders) | 2 | 1
Myocardial infarction (Cardiac disorders) | 2 | 2
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 3 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Angle closure glaucoma (Eye disorders) | 1 | 0
Retinal vein occlusion (Eye disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal incarcerated hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Colitis microscopic (Gastrointestinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 6
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 2 | 0
Chronic fatigue syndrome (General disorders) | 1 | 0
Impaired healing (General disorders) | 0 | 1
Pneumatosis (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 0
Sudden cardiac death (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic cyst (Hepatobiliary disorders) | 1 | 0
Chronic allograft nephropathy (Immune system disorders) | 1 | 2
Kidney transplant rejection (Immune system disorders) | 19 | 7
Renal transplant failure (Immune system disorders) | 0 | 1
Anal abscess (Infections and infestations) | 1 | 0
BK virus infection (Infections and infestations) | 1 | 2
Bacterial pyelonephritis (Infections and infestations) | 3 | 0
Bronchitis (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 1 | 3
Chronic sinusitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 2
Diverticulitis (Infections and infestations) | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Escherichia infection (Infections and infestations) | 1 | 0
Escherichia sepsis (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 6
Gastroenteritis norovirus (Infections and infestations) | 1 | 1
Gastroenteritis rotavirus (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Hepatic cyst infection (Infections and infestations) | 1 | 1
Herpes zoster (Infections and infestations) | 2 | 0
Histoplasmosis disseminated (Infections and infestations) | 0 | 1
Infected cyst (Infections and infestations) | 1 | 0
Infected lymphocele (Infections and infestations) | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 2 | 2
Localised infection (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Necrotising soft tissue infection (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 5 | 7
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 1 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 1
Renal cyst infection (Infections and infestations) | 0 | 2
Renal graft infection (Infections and infestations) | 2 | 1
Sepsis (Infections and infestations) | 4 | 2
Subcutaneous abscess (Infections and infestations) | 0 | 1
Systemic candida (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 7 | 7
Urosepsis (Infections and infestations) | 6 | 3
Wound infection (Infections and infestations) | 1 | 2
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1 | 2
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 2 | 0
Post procedural fever (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Shunt blood flow excessive (Injury, poisoning and procedural complications) | 1 | 0
Shunt occlusion (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 1
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 2 | 2
Donor specific antibody present (Investigations) | 1 | 0
Norovirus test positive (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Steroid diabetes (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 2
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 5
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 5
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebral artery stenosis (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 3
Confusional state (Psychiatric disorders) | 1 | 0
Depressive delusion (Psychiatric disorders) | 0 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 4 | 5
Bladder diverticulum (Renal and urinary disorders) | 1 | 0
Glomerulonephritis (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 2 | 0
Renal artery stenosis (Renal and urinary disorders) | 0 | 1
Renal disorder (Renal and urinary disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Vesicoureteric reflux (Renal and urinary disorders) | 0 | 1
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Vulvar dysplasia (Reproductive system and breast disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 1
Dry gangrene (Vascular disorders) | 0 | 1
Extremity necrosis (Vascular disorders) | 2 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Hypotension (Vascular disorders) | 2 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 2
Peripheral artery stenosis (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Belatacept (N=221) | CNI-Based Regimen (N=222)
Abdominal pain (Gastrointestinal disorders) | 12 | 13
Diarrhoea (Gastrointestinal disorders) | 47 | 61
Nausea (Gastrointestinal disorders) | 15 | 11
Vomiting (Gastrointestinal disorders) | 10 | 13
Fatigue (General disorders) | 22 | 15
Oedema peripheral (General disorders) | 22 | 35
Pyrexia (General disorders) | 20 | 17
Bronchitis (Infections and infestations) | 23 | 18
Nasopharyngitis (Infections and infestations) | 44 | 50
Upper respiratory tract infection (Infections and infestations) | 17 | 18
Urinary tract infection (Infections and infestations) | 37 | 33
Blood creatinine increased (Investigations) | 20 | 18
Arthralgia (Musculoskeletal and connective tissue disorders) | 21 | 23
Back pain (Musculoskeletal and connective tissue disorders) | 18 | 22
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 20
Dizziness (Nervous system disorders) | 15 | 8
Headache (Nervous system disorders) | 27 | 23
Tremor (Nervous system disorders) | 6 | 12
Insomnia (Psychiatric disorders) | 9 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 31 | 20
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 12
Hypertension (Vascular disorders) | 29 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/72/NCT01820572/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-21): https://cdn.clinicaltrials.gov/large-docs/72/NCT01820572/SAP_001.pdf